CLINICAL TRIAL: NCT04824469
Title: The Effects of Web-Based Training and Telephone Follow-up Developed for Covid-19 Patients on Symptom Management, Medication Compliance and Quality of Life
Brief Title: The Effects of Web-Based Training for Covid-19 Patients on Symptom Management, Medication Compliance and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ebru Arslan Özdemir, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EkisehirOsmangaziU
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: web based consulting; Medication Compliance; symptom management; covid-19; life quality
MeSH Terms: conditions — COVID-19; Medication Adherence

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web based training (Experimental): * Patients on the first day; Patient Information Form (1st and 2nd part), Memorial Symptom Assessment Scale, Covid-19 Symptom Assessment Inventory, Morisky Compliance Scale, World Health Organization Quality of Life Scale Short Form Turkish Version, E-Health literacy scale on website or mobile devices Google via the form or by sending a phone link.
  * Morisky Compliance Scale will be applied on the 7th day by sending a link to the website or mobile devices via google form.
  * Patients in the intervention group will be asked to fill out the Covid-19 Symptom Assessment Inventory on the website when they experience changes in their symptoms.
  * Patients in the intervention group will be provided with web-based training and telephone (SMS) reminder service for 4 weeks.
  * All questionnaires and web site evaluation form will be filled in the pre-test after 4 weeks.
  Interventions: Other: intervention group
- standard care (No Intervention): The scales applied to the intervention group on the first day, by sending the E-Health literacy scale form or phone link via Google on mobile devices. The symptoms of the patients in the control group will be evaluated at the end of the 1st day, 7th day, 14th day and 4th day. No intervention was planned for the patients in the control group during the follow-up. In the standard practice protocol, after patients are informed for follow-up and treatment at home, they are called by the Ministry of Health and family physicians for symptom follow-up. The standard hospital protocol does not include a scheduled training program, telephone monitoring, or web-based training. After collecting the data in the intervention group, the website will be opened to the use of the control group.

INTERVENTIONS:
Other: intervention group — web based training: By establishing a website, training on drug use, symptom management and quality of life will be provided.
  Arms: web based training

SUMMARY:
2019 coronavirus disease (Covid-19) is a virus that emerged in Wuhan, China in late 2019, spread all over the world in a short time and causes severe acute respiratory syndrome and pneumonia. The World Health Organization classified the COVID-19 outbreak as an "international public health emergency" on January 30 and declared a global epidemic (pandemic) on March 11, 2020, due to the rapid spread of the virus all over the world. speed in the number of cases and deaths. Covidien-19 first cases were reported in Turkey on 10 March 2020 and the number of cases has risen steadily.

The total number of COVID-19 cases worldwide on 31.01.2021; It was reported to be 101,917,147 and the total number of deaths was 2,205,515 (https://covid19.who.int/).

Considering that the number of cases is constantly increasing, it is obvious that hospitals will not meet the entire epidemic burden. During this period, home care has emerged as an alternative way to effectively alleviate the epidemic burden. Home healthcare during the COVID-19 pandemic; Four roles have stood out: home diagnosis, follow-up, treatment, and care.

Protective measures for home isolation of Covid-19 patients are the current method used to prevent the spread of cases. Possible or definite cases that do not have an indication for hospitalization, have a mild clinic and do not accompany severe chronic disease that may lead to a severe course of covid-19 are followed at home until their symptoms improve. In addition, patients who are hospitalized and meet discharge criteria can complete their recovery processes at home. Isolation is terminated on the 14th day at the earliest following the improvement of symptoms in patients who are followed at home. Reducing the contact of people, isolating certain and suspicious cases and effective use of personal protective equipment play an important role in combating the epidemic. It is thought that the training that COVID-19 cases to be followed up and treated at home will be effective in drug compliance, symptom management and quality of life will be effective in the management of the disease.

1251 / 5000 Çeviri sonuçları The universe of the research will be composed of people who apply to Zonguldak Atatürk State Hospital Emergency Service and Covid-19 Polyclinics. . The sample of the study, who accepted to participate in the study, was diagnosed with Covid-19 with U07.3 ICD code according to the results of PCR (Polymerase Chain Reaction) test and Thorax CT (Thorax CT), and was recommended to be followed up and treated at home by the Zonguldak Public Health Department It is planned to create individuals who meet the criteria.

DETAILED DESCRIPTION:
G power analysis program was used to determine the sample size. The research will be conducted in two groups, an intervention and a control group. With professional support in calculating the sample size of the study, the sample size calculated at a 5% margin of error and a 95% confidence interval was found to be 128. However, against the possibility of sample losses during the follow-up process, the individual diagnosed with Covid-19 will be added to the number of samples by adding 20% (13 participants will be added for each group. 77 interventions in total, 77 controls) will be included in the study. Participants who meet the inclusion criteria and agree to participate in the study will be randomly assigned to the intervention and control groups.

DATA COLLECTION TOOLS

* Patient information form
* Memorial Symptom Rating Scale
* Covid-19 Symptom Assessment Inventory
* Morisky Adaptation Scale (Muö)
* World Health Organization Quality of Life Inventory Short Form Turkish Version
* E-Health literacy scale
* Opinion Form Regarding the Web Based Training Program
* DISCERN Guide (Expert Opinions)
* Website Content Evaluation Form (Expert Opinions)

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18,
* Does not have a communication problem that prevents participation in research or education, such as inability to understand / speak Turkish,
* Being literate,
* Residing in Zonguldak province, applying to hospitals in the province and diagnosed with Covid-19 according to PCR (Polymerase Chain Reaction) test and Thorax CT (Thorax computed tomography) results by the radiation teams and deemed appropriate for home follow-up by the Zonguldak Public Health Directorate,
* Having active Internet access and actively using a computer / tablet or smartphone,
* Patients who agree to participate in the study

Exclusion Criteria:

* No internet connection at home or on the phone,
* Do not know how to use internet and computers,
* Having a communication problem that prevents participation in research or education, such as inability to understand / speak Turkish, Patients who were previously diagnosed with Covid-19 and treated at home or in hospital,
* With severe insufficiency (Heart failure, Kidney failure, Immune system failure)
* Illiterate individuals will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pre-intervention measurements | first day
  The Covid-19 symptom assessment inventory prepared by scanning the literature will be used to monitor the symptoms. The high score obtained from the inventory indicates the need for disease management.
Pre-intervention measurements | first day
  Morisky drug compliance scale to measure drug compliance: is a self-report scale consisting of four questions. The questions are answered as "yes (1 point) and no (0 point). Increasing the score obtained from the scale indicates that drug compliance is low.
Pre-intervention measurements | first day
  The Turkish version of the World Health Organization Quality of Life Inventory Short Form will be used to measure the quality of life. The scale is a Likert type form consisting of 27 questions. Higher total scores obtained from the scale indicate a good quality of life.

SECONDARY OUTCOMES:
Post-intervention measurements | 1. month
  The Covid-19 symptom assessment inventory prepared by scanning the literature will be used to monitor symptoms. The high score obtained from the inventory indicates that the need for disease management continues.
Post-intervention measurements | 1. week
  Morisky drug compliance scale to measure drug compliance: is a self-report scale consisting of four questions. The questions are answered as "yes (1 point) and no (0 point). Increasing the score obtained from the scale indicates that drug compliance is low.
Post-intervention measurements | 1. month
  The Turkish version of the World Health Organization Quality of Life Inventory Short Form will be used to measure the quality of life. The scale is a Likert type form consisting of 27 questions. Higher total scores obtained from the scale indicate a good quality of life.

IPD SHARING:
Plan to Share IPD: No